CLINICAL TRIAL: NCT07325513
Title: Machine Learning in Guiding rTMS Treatment for GWI-Related Headaches and Body Pain
Acronym: SVM - GWI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H2500180
Record Dates: First submitted 2026-01-06; First posted 2026-01-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Gulf War Illness; Headache; Muscle and Joint Pain
Keywords: Repetitive Transcranial Magnetic Stimulation (rTMS); Support Vector Machine (SVM); Headache; Machine Learning; Muscle and Joint Pain
MeSH Terms: conditions — Headache; Arthralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Group A: Predicted Respondent at LDLPFC (Active Comparator)
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation
- Group B: Predicted Non-respondent at LDLPFC (Active Comparator)
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation
- Group C: Predicted Respondent at LDLPFC and LMC (Active Comparator)
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation
- Group D: Predicted Non-respondent at LDLPFC and LMC (Active Comparator)
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Active Repetitive Transcranial Magnetic Stimulation — rTMS will be administered to the LDLPFC with an active coil.
  Arms: Group A: Predicted Respondent at LDLPFC
Device: Active Repetitive Transcranial Magnetic Stimulation — rTMS will be administered to the LDLPFC with an active coil.
  Arms: Group B: Predicted Non-respondent at LDLPFC
Device: Active Repetitive Transcranial Magnetic Stimulation — rTMS will be administered to the LDLPFC and LMC with an active coil.
  Arms: Group C: Predicted Respondent at LDLPFC and LMC
Device: Active Repetitive Transcranial Magnetic Stimulation — rTMS will be administered to the LDLPFC and LMC with an active coil.
  Arms: Group D: Predicted Non-respondent at LDLPFC and LMC

SUMMARY:
The goal of this clinical trial is to create a machine learning algorithm to improve active repetitive transcranial magnetic stimulation (rTMS) treatments for veterans and/or active military personnel by alleviating Gulf War Illness related headaches and body pain (GWI-HAP). This study aims to develop and validate a Support Vector Machine (SVM) model that could replace the trial-and-error process by assessing functional connectivity provided by resting state functional magnetic resonance imaging (rs-fMRI) data to predict the most effective rTMS protocol for each person. All participants will be receiving active rTMS treatment.

The main questions it intends to answer are:

1. Does the SVM model predict a more effective treatment response rate for predicted respondents undergoing active rTMS at the left dorsolateral prefrontal cortex (DLPFC) compared to predicted non-respondents?
2. Does the SVM model predict a more effective treatment response rate while undergoing active rTMS at the left dorsolateral prefrontal cortex (DLPFC) and left motor cortex (LMC) in predicted respondents compared to predicted non-respondents?

Participants will undergo the following:

1. Receive a total of 13 active rTMS treatment sessions over 3-4 months.
2. Visit the clinic for a total of 15 visits for assessments, check ups, and treatments.
3. Keep a daily log of their headaches, muscle and joint pain throughout the study.

DETAILED DESCRIPTION:
This study aims to enroll a total of 140 veterans and/or active military personnel over the 4-year study period at the VA San Diego Healthcare System (VASDHS). Participants will be randomized into receiving treatments at the left DLPFC or left DLPFC and LMC, then placed into predicted respondent or non-respondent groups. They will be assigned to 1 of 4 groups:

Group A: Predicted Respondent at Left DLPFC Group B: Predicted Non-respondent at Left DLPFC Group C: Predicted Respondent at Left DLPFC and LMC Group D: Predicted Non-respondent at Left DLPFC and LMC

Participation in this study will require 15 total visits to the VASDHS over the course of 3-4 months. The visits will be separated in the following phases:

1. Pre-Treatment Assessments Phase (Weeks 1-2): Visit 1 (Screening) and Visit 2 (Baseline Assessments)
2. Induction Treatment Phase (Weeks 2-4): Visits 3-12 (Weekday active rTMS sessions at >24 hours and <72 hours apart)
3. Follow-Up and Maintenance Phase (Weeks 5-10): Visit 13 (1 week follow-up); Visit 14 (1 month follow-up); Visit 15 (2 months follow-up); All maintenance visits follow the final treatment of the induction phase.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Veteran or active military personnel
* Between the ages of 18 and 65 years old
* Served in the Persian Gulf region for at least 30 consecutive days between August 1, 1990, and July 31, 1991
* Meets the CDC Criteria for GWVI (GWI), with symptoms starting during or after the 1990-1991 Persian Gulf deployment. Symptoms must be present for at least 6 months prior to enrollment in the study. Symptoms must be present in at least 2 of the 3 categories of fatigue, musculoskeletal, and mood cognitive.
* Meets the Kansas Criteria for GWVI (GWI), with symptoms starting during or after the 1990-1991 Persian Gulf deployment. Symptoms must be present for at least 6 months prior to enrollment in the study. Qualifying symptoms must be at least moderate in severity and/or multiple symptoms must be present within at least 3 of 6 categories consisting of fatigue/sleep, neurological/cognitive/mood, pain, respiratory, gastroenterological, and dermatological symptomology.
* Average Overall Daily Muscle Pain Intensity ≥3 on a 0-10 NPRS, present for at least 6 months
* Average Overall Daily Extremities Joint Pain Intensity ≥3 on a 0-10 NPRS, present for at least 6 months
* Average Headache Exacerbation Intensity ≥3 on a 0-10 NPRS, with headaches occurring for at least 6 months
* Headache Exacerbation/attack ≥ 1 time per week with the average intensity ≥3 on a 0-10 NPS, lasting > 1 hour in the past three months
* International Headache Society Criteria for Migraine Headache without aura

Exclusion Criteria:

* Children under the age of 18
* Pregnant women
* Individuals with cognitive/decisional impairment
* Non-English speaking individuals
* Prisoners of War
* Incarcerated individuals
* VA employees - including VA paid, IPA, or WOC
* Students of the institution or of the investigator
* Patients with cancer
* History of pacemaker implant
* Presence of ferromagnetic material (e.g., bullet fragment, shrapnel, device implant) in the brain or body that will prohibit the patients from having a brain MRI
* History of dementia, major psychiatric diseases, or life-threatening diseases
* Presence of any other chronic neuropathic pain states such as Complex Regional Pain Syndrome or Painful Peripheral Neuropathy
* Known diagnosis of moderate to severe osteoarthritis and/or rheumatologic joint pain prior to the GWI deployment
* Low back pain with mechanical origins such as lumbar radiculopathy or radiculitis or lumbar facet arthropathy
* Concurrent conditions, like lupus, that can produce symptoms compatible with GWVI
* History of seizure
* Pending litigation
* History of Traumatic Brain Injury-related headaches
* Chronic Tension or Cluster Headache. However, subjects with occasional tension headaches (less than once every three months and lasting no more than 24 hours) will not be excluded from the study.
* Ongoing Cognitive Rehabilitation or Treatment of PTSD
* Recent exacerbation of anxiety disorder symptoms, active substance dependence, and/or current psychotic symptoms
* Ongoing suicidal/homicidal ideation or recent (in the past 6 months) suicidal attempts
* Patients who receive any narcotic-based analgesic, topical analgesics over the affected site, steroid and local anesthetic injection, anticonvulsants, and antipsychotic medications less than 7 days prior to the pretreatment assessment
* Patients who do not agree to avoid use of non-pharmacologic treatments, including but not limited to, transcutaneous electrical nerve stimulation unit (TENS), acupuncture, acupressure, and therapeutic massage during the entire study.
* Patients who do not agree to use additional acetaminophen (up to a maximum total of 3g per day) as the only rescue medication
* Patients who have received rTMS within the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity - Mechanical Visual Analogue Scale (M-VAS) | From baseline to the end of treatment at 16 weeks
  A scale that ranges from 0 to 10 ("No pain" to "Worst possible pain").
Headache and Pain Log | From enrollment to the end of treatment at 16 weeks
  A personal daily log is used to track the subject's headaches, muscle and joint pain throughout the course of the study based on a range of 0 to 10, with higher scores indicating more severe pain.
Mood - Hamilton Rating Scale for Depression (HRSD) | From baseline to end of treatment at 16 weeks
  This scale is a well-established questionnaire which consists of twenty-one questions and rates the severity of symptoms observed in depression such as low mood, insomnia, agitation, anxiety and weight loss. Only the first 17 items are used for the overall scoring. A score between 14 and 18 represents a moderate form of depression and a score greater than 19 represents severe depression.
Pain Severity - Brief Pain Inventory-Short Form (BPI-sf) | Baseline, 1-week, 1-month, 2-months
  This is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during the 24-hour period prior to evaluation. The BPI-sf consists of five questions. Four items measure pain on 11-point response scales from 0 to 10 ("No Pain" to "Pain as bad as you can imagine"). Another item, containing 7 sub-questions, evaluates the level of pain interference with daily functioning on 11-point response scales from 0 to 10 ("Does not interfere" to "Completely interferes"). Items 3-6 are summed together for a total average pain severity score.
Pain Severity - Brief Pain Inventory-Short Form (BPI-sf) | Baseline, 1-week, 1-month, 2-months
  This is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during the 24-hour period prior to evaluation. The BPI-sf consists of five questions. Four items measure pain on 11-point response scales from 0 to 10 ("No Pain" to "Pain as bad as you can imagine"). Another item, containing 7 sub-questions, evaluates the level of pain interference with daily functioning on 11-point response scales from 0 to 10 ("Does not interfere" to "Completely interferes"). Items 9A-9G are summed together for a total pain interference score.
Pain Quality and Intensity - Short Form McGill Pain Questionnaire (SF-MPQ) | Baseline, 1-week, 1-month, 2-months
  This is a self-report questionnaire that allows individuals to describe the quality and intensity of pain they are experiencing. This will be used to assess the sensory and affective aspects of muscle pain. The SF-MPQ consists of fifteen questions; items 1-11 are measured on a 4-point response scale ranging from 0 to 3 ("None" to "Severe"). Items 12-15 include a visual analogue scale (VAS) from "No pain" to "Worst possible pain" and Present Pain Intensity (PPI) ranging from 0 to 5 ("No pain" to "Excruciating") ranking overall pain intensity for a total average muscle pain score. This is calculated via the average VAS scores (0-100) with 0 indicating no pain and 100 equivalent to the worst pain possible.
Pain Quality and Intensity - Short Form McGill Pain Questionnaire (SF-MPQ) | Baseline, 1-week, 1-month, 2-months
  This is a self-report questionnaire that allows individuals to describe the quality and intensity of pain they are experiencing. This will be used to assess the sensory and affective aspects of joint pain. The SF-MPQ consists of fifteen questions; items 1-11 are measured on a 4-point response scale ranging from 0 to 3 ("None" to "Severe"). Items 12-15 include a visual analogue scale (VAS) from "No pain" to "Worst possible pain" and Present Pain Intensity (PPI) ranging from 0 to 5 ("No pain" to "Excruciating") ranking overall pain intensity for a total average joint pain score. This is calculated via the average VAS scores (0-100) with 0 indicating no pain and 100 equivalent to the worst pain possible.
Functionality - Revised Fibromyalgia Impact Questionnaire | Baseline, 1-week, 1-month, 2-months
  A questionnaire to evaluate the function, overall impact and symptoms of Fibromyalgia. The 3 categories are calculated by the sum of the scores to produce a total score. Each item ranges from 0-10 and the total score is 0-100 with high scores indicating more severe impact.
Pain Intensity - New Clinical Fibromyalgia Diagnostic Criteria - Part 1 | Baseline, 1-week, 1-month, 2-months
  Patients will be asked to rate the average (over the past week) intensity of muscle pain up to 12 locations of the body. This is calculated by the Widespread Pain Index (WPI) total score ranging from 0 to 19 and a marker visual analogue scale (MVAS) ranging from 0 to 100.
Pain Severity - Headache Impact Test (HIT-6) | Baseline, 1-week, 1-month, 2-months
  This test measures how impact headaches affect the individual's ability to function in different domains. This six question test evaluates the severity of headache pain from "Never" to "Always" with a total range between 36-78, higher scores indicating greater impact on functionality.
Pain Severity - Neurobehavioral Symptoms Inventory (NSI) | Baseline, 1-week, 1-month, 2-months
  This twenty-two self-report questionnaire on the severity of each symptom is measured using a 5-point response scale ranging from 0 to 4 ("None - Rarely if ever present; not a problem at all" to "Very Severe - Almost always present and I have been unable to perform at work, school or home due to this problem; I probably cannot function without help"). It asks the subjects to indicate the extent to which each symptom has disturbed them. The total score ranges from 0 to 88 with a higher score indicating very severe symptom disruption.
Sleep Quality - Pittsburgh Sleep Quality Index (PSQI) | Baseline, 1-week, 1-month, 2-months
  This index has nineteen individual items which are used to generate 7 composite scores on: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The 7 components measure sleep habits and sum together to measure global sleep quality with a high score of 0-21 with a higher score indicating worse sleep quality.
Sleep Severity - Insomnia Severity Index | Baseline, 1-week, 1-month, 2-months
  This index consists of seven questions that depict the severity of sleep difficulties within the past 2 weeks on a 5-point response scale that rates satisfaction, noticeability, distress, and interference with daily functioning. A score between 15 and 21 suggests moderately severe clinical insomnia. A score of 22 or greater represents severe clinical insomnia.
Quality of Life - Veteran RAND 36-item Health Survey (VR-36+PCS and MCS) | Baseline, 1-week, 1-month, 2-months
  A patient-reported survey of patient health. It is a measure of health status and quality of life in regards to eight main areas: vitality, physical functioning, bodily pain, health perceptions, physical, emotional, and social role functioning and mental health.
Multidimensional Fatigue Inventory | Baseline, 1-week, 1-month, 2-months
  A twenty item self-report instrument with 4 categories total designed to measure fatigue level (24-96) with a higher score indicating more severe fatigue.
Chronic Fatigue Severity Scale | Baseline, 1-week, 1-month, 2-months
  A Likert scale consisting of nine items that assess fatigue severity and functionality. The sum of all questions provides total fatigue level 8-63 with a higher score being more severe. A score over 36 indicates patient may be suffering from fatigue.

SECONDARY OUTCOMES:
Opiate/Medication Assessment | From the baseline to the end of treatment at 16 weeks
  This assessment evaluates opiate consumption over the duration of the study. Opioids and narcotics are converted to their morphine equivalent value on a daily basis. Values during each measurement period are added up and divided by the number of weeks to determine weekly usage.

IPD SHARING:
Plan to Share IPD: No